CLINICAL TRIAL: NCT05400083
Title: Prevention of Incisional Hernia With Biosynthetic Mesh at the Site of Temporary Ileostomy Closure
Brief Title: Prevention of Incisional Hernia With Biosynthetic Mesh at the Site of Temporary Ileostomy Closure (PRINCESS)
Acronym: PRINCESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Umberto Bracale, Prof., Federico II University
Other Study IDs: 471/20
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prophylactic mesh reinforcement of the abdominal wall at the site of temporary ileostomy closure is effective in preventing postoperative incisional hernia.

This prospective, multicenter, observational study will evaluate performance of Phasix biosynthetic mesh when used to reinforce fascial closure .

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be informed about the study, and will have read; understood and signed the informed consent
* Subjects of either gender that are at least the age of 18 years
* Subjects will be undergoing ileostomy reversal with retromuscular placement technique of the Phasix biosynthetic mesh reinforcement

Exclusion Criteria:

* Subjects who, in the surgeon's opinion, would have a difficult time comprehending or complying with the requirements of the study
* Subjects with parastomal hernia or midline incisional hernia
* Subjects who required midline laparotomy during ileostomy reversal

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: General and teaching hospitals
Sampling Method: Non-Probability Sample
Enrollment: 203 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia rate | at 24 months
  CT scan or Ultrasound as imaging to detect incisional hernia

SECONDARY OUTCOMES:
Early and Long-term Complication Rates | after surgery to 24 months
  Clavien-Dindo classification
Postoperative pain | after surgery to 24 months
  Visual analogue scales (VAS) Range: 1-100. Higher score correlates with more pain
Quality of life by Carolinas Comfort Scale (CCS) and Euro-Qol 5D-5L questionnaires | after surgery to 24 months
  CCS - Range: 0-115. Higher score correlates with worse outcome
Budget Impact Analysis | after surgery to 24 months
  Healthcare Cost Analysis including direct costs (fixed and variable)

CONTACTS AND LOCATIONS:
Locations (1):
- Minimally Invasive General and Oncologic Surgery Unit - Univesity of Naples Federico II, Naples, Italy